CLINICAL TRIAL: NCT03211949
Title: Topographic Assessment of the Medial Antebrachial Cutaneous Nerve Variations at the Axilla and Above the Cubital Fossa Using Ultrasonography
Brief Title: Ultrasound Guided Topographic Mapping of Medial Antebrachial Cutaneous Nerve
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, Dr M. B. Breebaart, md, University Hospital, Antwerp
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 14/41/427
Record Dates: First submitted 2014-10-30; First posted 2017-07-11 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Nerve Block; Surgery; Anesthesia; Brachial Plexus Block
Keywords: axillary nerve block
MeSH Terms: interventions — Mepivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- axillary block with infiltration MCAN (Experimental): With the performance of the axillary blok, 2 ml of scandicaine will be placed around the medial cutaneous ante brachial nerve (MACN)
  Interventions: Procedure: axillary block; Drug: Scandicaine

INTERVENTIONS:
Procedure: axillary block — 2 ml of scandicaine 1.5 % is deposited in an inplane technique around the medial antebrachial cutaneous nerve with a 22 G sonoplex needle as a surplus to an axillary block
Drug: Scandicaine — 2 ml of scandicaine 1.5 % is deposited in an inplane technique around the medial antebrachial cutaneous nerve with a 22 G sonoplex needle as a surplus to an axillary block
  Other Names: mepivacaine

SUMMARY:
Blocking the medial antebrachial cutaneous nerve (MACN) during an axillary block often a subcutaneous wheal of local anesthetics is made what is described as painful. With the improvement of the resolution of the ultrasound machines smaller structures and nerves can be visable. In this study topographic assessment will made of the anatomical variation of the medial antebrachial cutaneous nerve (MACN) by ultrasound in the axilla and 5 cm above the cubital fossa of the arm.

DETAILED DESCRIPTION:
The ethics committee will approved the study and informed consent is obtained. Patients with contraindications for regional anaesthesia will be excluded from the study. 150 patients will be included The arm is placed above and beside the head for scanning (abduction 90 degrees at the shoulder and 90 degrees flexion at the elbow with external rotation) Ultrasound is performed with a 12-18 MHz (Mega-Herz) linear probe (BK medical). The frequency is set to 18 MHz and the depth to 3 cm and adjusted to 1 cm below the brachial artery .

The terminal nerves of the brachial plexus (median, ulnar,radial an d musculocutaneous) are identified at the axillary fossa in a routine fashion described by Ranganath (see references).

After identifying the MACN at the axilla and 5 cm above the cubital fossa, the images at these two sites will be stored after digital marking of the MACN, the medial and ulnar nerve and the and radial nerve on the frozen ultrasound image. Its position relative to the venous structure and the artery at the axilla will be registered in the axilla at the lower border of the conjoint tendon of the teres major and the latissimus dorsi muscle.

After scanning the skin will be prepared with an aseptic solution and an axillary block will be performed with a 55 mm sonoplex 22 G short bevel ultrasound needle (Pajunk). With a partly in plane (ulnar, radial and MACN) and partly out of plane (median & musculocutaneous nerve) technique . Mepivacaine 1.5 % will be injected around each nerve in the following order: Ulnar nerve, MACN, radial nerve, median nerve and musculocutaneous nerve. The time at which the MACN is blocked will be noted. For each nerve 5 ml of local anaesthetic solution will be injected except for the MACN nerve where 3 ml will be used because of its smaller caliber.

Nerve stimulation will be used with a current of 0,2 mA (milli Amps). Following completion of the block the dermatome supplied by the MACN will be tested by loss of cold sensation. After 20 minutes the dermatomes and motor function of all nerves are tested by elbow flexion and extension, primarily thumb opposition and abduction of the index finger. Sensory block is tested at the fifth finger (ulnar nerve, the hand palm at the thumb (medial nerve)and the dorsum of the hand ( radial nerve), the lateral (musculocutaneous nerve) and medial skin ( MACN) of the forearm.

Skin will be prepared with an aseptic solution and an axillary block will be performed with deposition of local anesthetic around the MACN.

Data processing. The locations of the different nerves will be displayed in a pie chart with the axillary artery in the centre, as well as the relative position to the basilic vein. Statistics will only be descriptive .

ELIGIBILITY:
Inclusion Criteria:

* all patients scheduled for lower arm/hand surgery

Exclusion Criteria:

* patient refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2014-09; Primary Completion 2019-12 (Actual); Study Completion 2020-01-30 (Actual)

PRIMARY OUTCOMES:
anatomical mapping of the MACN relative to the basilic vein, radial nerve and ulnar nerve | up to 30 minutes
  an ultrasound image will be stored with the structures marked

CONTACTS AND LOCATIONS:
Overall Officials: margaretha breebaart, Principal Investigator — Univeristy Hospital Antwerp
Locations (1):
- University Hospital Antwerp, Antwerp, Belgium

REFERENCES:
- [Background] Ranganath A, Srinivasan KK, Iohom G. Ultrasound guided axillary brachial plexus block. Med Ultrason. 2014 Sep;16(3):246-51. doi: 10.11152/mu.2013.2066.163.2kks. PMID 25110766